CLINICAL TRIAL: NCT02990351
Title: Loco-regional Treatment for HCC Patients
Brief Title: Efficacy of Loco-regional Treatment for Hepatocellular Carcinoma Prior to Living Donor Liver Transplantation in Egypt
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Iman Fawzy Montasser, Associate profesor of tropical medicine , Ain Shams university, Ain Shams University
Other Study IDs: HCC and liver transplantation
Record Dates: First submitted 2016-12-04; First posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Hepatocellular Carcinoma (HCC); Living Donor Liver Transplantation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HCC patients: 29 HCC patients who had loco regional therapies for HCC were analyzed. Twenty patients met the Milan criteria (68.97%) & 4 (13.8%) were beyond Milan but met UCSF criteria and 5 were exceeding UCSF criteria (17.2%).All patients underwent preoperative LRTs, The protocol of bridging/down staging, methods, duration of follow up, the number of the patients who were successfully down-staged before LT and their outcomes after LT were recorded.
  Interventions: Procedure: loco regional therapies for HCC

INTERVENTIONS:
Procedure: loco regional therapies for HCC — 29 HCC patients received locoregonal therapy as a bridging therapy for those who were within milan and as downstaging for those were initially beyond milan. The main LRT types used for our patients were TACE and or RFA and microwave ablation

SUMMARY:
This study aimed to analyze the outcomes of loco-regional treatment prior Living Donor Liver Transplantation in patients with HCC.

DETAILED DESCRIPTION:
50 patients received LDLT at Ain Shams Centre for Organ Transplantation (ASCOT) over 1 year of whom data of 29 HCC patients were analyzed. Twenty patients met the Milan criteria (68.97%) & 4 (13.8%) were beyond Milan but met UCSF criteria and 5 were exceeding UCSF criteria (17.2%).All patients underwent preoperative LRTs, The protocol of bridging/down staging, methods, duration of follow up, the number of the patients who were successfully down-staged before LT and their outcomes after LT were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients 18-65 years
2. Patients transplanted for HCC within Milan and UCSF criteria who underwent pre transplant bridge or down staging treatment for HCC

Exclusion Criteria:

1. Tumor progression on the waiting list
2. Vascular invasion by imaging studies
3. Extrahepatic or lymph node metastasis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Egyptian patients prepared for living donor liver transplantation , at Ain Shams Centre for Organ Transplantation (ASCOT) , Cairo Egypt
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Radiological Response ( complete / partial / tumour progression)in the Radiology (CT/ MRI) before transplantation | 3 months
  the success of loco-regional therapy for hepatocellular carcinoma in term of radiological complete or partial response in the last spiral triphasic abdominal CT and /or MRI before transpalantation

SECONDARY OUTCOMES:
the degree of accuracy between the last CT/ MRI and the pathology of explant in term of number , size and ablation (complete necrosis ) for HCC | 3 months
  1. presence of viable tumour tissue in the explant pathology,
  2. mictro vascular invasion
  3. capsular or lymph node invasion the degree of accuracy between the last CT/ MRI and the pathology of explant

IPD SHARING:
Plan to Share IPD: Undecided